CLINICAL TRIAL: NCT02375139
Title: A Randomized, Open-label, Crossover, Single Dose Clinical Trial to Investigate Safety/Tolerability and Pharmacokinetics of DA-1229_01 (Evogliptin/Metformin XR 2.5/500 mg x 2 Tablets) Compared to Co-administration of Evogliptin 5 mg and Metformin XR 1000 mg After Single Oral Administration in Healthy Male Volunteers
Brief Title: A Clinical Trial to Investigate Safety/Tolerability and Pharmacokinetics of DA-1229_01(Evogliptin/Metformin XR 2.5/500 mg x 2 Tablets) Compared to Co-administration of Evogliptin 5 mg and Metformin XR 1000 mg in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA-1229_01
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 4-(3-amino-4-(2,4,5-trifluorophenyl)butanoyl)-3-(tert-butoxymethyl)piperazin-2-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DA-1229_01 → E+M (Experimental): DA-1229_01 : Evogliptin/Metformin XR 2.5/500mg x 2 Tablets E : Evogliptin 5 mg M : Metformin XR 1000 mg
  Interventions: Drug: DA-1229_01; Drug: E+M
- E+M → DA-1229_01 (Experimental): DA-1229_01 : Evogliptin/Metformin XR 2.5/500mg x 2 Tablets E : Evogliptin 5 mg M : Metformin XR 1000 mg
  Interventions: Drug: DA-1229_01; Drug: E+M

INTERVENTIONS:
Drug: DA-1229_01 — complex single administration
  Other Names: Evogliptin/Metformin XR 2.5/500 mg x 2 Tablets
Drug: E+M — co-administration of 2 drugs
  Other Names: Evogliptin 5 mg + Metformin XR 1000 mg

SUMMARY:
This Phase I clinical study is to evaluate the safety/tolerability and pharmacokinetics of DA-1229_01(Evogliptin/Metformin XR 2.5/500 mg x 2 tablets).

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 60-125mg/dL glucose level(at screening)
* Volunteer who totally understands the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Volunteer who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology, immunology, pulmonary, endocrine, hematooncology, cardiology, mental disorder)
* Volunteer who had GI tract disease(Crohn's disease, ulcer, acute or chronic pancreatitis) or surgery(appendectomy, hernioplasty are excluded)
* Volunteer who had drug(Aspirin, antibiotics) hypersensitivity reaction
* Subject who already participated in other trials in 2 months
* Subject who had whole blood donation in 2 months, or component blood donation in 1 months or transfusion

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC)last of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose
Maximum of concentration (Cmax) of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose

SECONDARY OUTCOMES:
Time of maximum concentration(Tmax) of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose
Terminal half-life(t1/2) of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose
Apparent Clearance(CL/F) of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose
Area Under Curve(AUC)inf of Evogliptin and Metformin | 1d(15d) pre-dose, 1,2,3,4,5,6,7,8,10,12,15,24,36,48,60,72h post-dose
  AUCinf = AUC last + Clast/λz

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, Ph.D, M.B.A, Principal Investigator — Seoul National University Hospital
Locations (1):
- Clinical Trial Center, Seoul National University Hospital, Seoul, South Korea